CLINICAL TRIAL: NCT03459807
Title: BOLD: A Trial of Blood Pressure Lowering in Dialysis
Brief Title: Blood Pressure Lowering in Dialysis (BOLD) Trial
Acronym: BOLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Washington (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-20963; R21DK114213 (NIH)
Record Dates: First submitted 2018-02-06; First posted 2018-03-09 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Blood Pressure; End Stage Renal Disease on Dialysis (Diagnosis); Chronic Kidney Diseases; Chronic Kidney Disease Stage 5
Keywords: Blood pressure; Hemodialysis; End-stage-renal-disease; Chronic kidney disease
MeSH Terms: conditions — Disease; Renal Insufficiency, Chronic | interventions — Antihypertensive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Home systolic blood pressure (SBP) <140 mmHg (Experimental): Participants will be asked to take morning and evening blood pressures every two weeks on a non-dialysis day.
  Participants will be asked to transmit these measures to the study team at minimum every 2 weeks either via Bluetooth technology, a manual log, telephone call, text message, e-mail, or verbal communication.
  Assigned intervention will be dry weight adjustment and/or adjustment of standard anti-hypertensive medications.
  Interventions: Drug: Anti-Hypertensive medications; Procedure: Dry Weight Adjustment
- Pre-dialysis SBP <140 mmHg (Active Comparator): Blood pressures taken in the clinical setting at prior to start of dialysis treatment will be recorded.
  Assigned intervention will be dry weight adjustment and/or adjustment of standard anti-hypertensive medications.
  Interventions: Drug: Anti-Hypertensive medications; Procedure: Dry Weight Adjustment

INTERVENTIONS:
Drug: Anti-Hypertensive medications — Use of standard Anti-Hypertensive medications
  Other Names: anti-hypertensive
Procedure: Dry Weight Adjustment — The participant's target post-dialysis dry weight is adjusted

SUMMARY:
Blood pressure may be one of the most important modifiable risk factors for cardiovascular disease in patients with end-stage-renal-disease undergoing maintenance hemodialysis. Although a systolic blood pressure <140 mmHg treatment target has been recommended, there remains uncertainty on which blood pressure should be targeted, more specifically that measured in the dialysis unit or at home. Observational studies have reported a paradoxical U-shaped associated with dialysis unit (pre-dialysis) systolic blood pressure and cardiovascular events and death (where blood pressure below 140 mmHg is actually linked with poor outcomes). Conversely, the same studies have reported a linear association between higher home systolic blood pressure and worse clinical outcomes, where blood pressure below 140 mmHg is associated with better outcomes. This pilot clinical trial aims to address this important question.

DETAILED DESCRIPTION:
Blood Pressure Lowering in Dialysis (BOLD) is a pilot randomized controlled trial of 50 maintenance hemodialysis patients in San Francisco and Seattle to test whether targeting a home systolic blood pressure <140 mmHg (versus a pre-dialysis systolic blood pressure <140 mmHg) is feasible and safe. The study duration is 4 months and blood pressure targets will be achieved through dry weight adjustment and adjustment of standard anti-hypertensive therapies by the study team. The primary outcomes are focused on feasibility and safety. The home blood pressure treatment arm will also have the opportunity to utilize a blood pressure monitor with Bluetooth capabilities. The rates of utilization of mobile health technology in this population will also be assessed as an outcome. This pilot trial will provide key data to design a larger trial focused on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Undergoing in-center, thrice weekly hemodialysis for treatment of end-stage-renal-disease
3. Greater than 3 months since initiation of dialysis
4. Age 18 years or above
5. Able to obtain a brachial blood pressure at dialysis and at home

Exclusion Criteria:

1. Pregnancy, anticipated pregnancy, or breastfeeding as this will require increase to more than three time a week dialysis and/or preclude use of some classes of blood pressure medications
2. Incarceration or institutionalized living which may prohibit measurement of home blood pressure
3. Participation in another intervention study that may affect blood pressure
4. Patients in whom systolic blood pressure is not measurable (e.g. those with left ventricular assist devices)
5. Hypotension: average pre-dialysis systolic blood pressure <100 mmHg over last 2 weeks prior to screening while not taking any blood pressure medications
6. Life expectancy <4 months
7. Anticipated living donor kidney transplant within 4 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-yuan Hsu, MD, Principal Investigator — Professor; Nisha Bansal, MD, MAS, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - UCSF, San Francisco, California
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] Flack JM, Neaton J, Grimm R Jr, Shih J, Cutler J, Ensrud K, MacMahon S. Blood pressure and mortality among men with prior myocardial infarction. Multiple Risk Factor Intervention Trial Research Group. Circulation. 1995 Nov 1;92(9):2437-45. doi: 10.1161/01.cir.92.9.2437. PMID 7586343
- [Background] MacMahon S, Peto R, Cutler J, Collins R, Sorlie P, Neaton J, Abbott R, Godwin J, Dyer A, Stamler J. Blood pressure, stroke, and coronary heart disease. Part 1, Prolonged differences in blood pressure: prospective observational studies corrected for the regression dilution bias. Lancet. 1990 Mar 31;335(8692):765-74. doi: 10.1016/0140-6736(90)90878-9. PMID 1969518
- [Background] Vamos EP, Harris M, Millett C, Pape UJ, Khunti K, Curcin V, Molokhia M, Majeed A. Association of systolic and diastolic blood pressure and all cause mortality in people with newly diagnosed type 2 diabetes: retrospective cohort study. BMJ. 2012 Aug 30;345:e5567. doi: 10.1136/bmj.e5567. PMID 22936794
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Sarnak MJ, Levey AS, Schoolwerth AC, Coresh J, Culleton B, Hamm LL, McCullough PA, Kasiske BL, Kelepouris E, Klag MJ, Parfrey P, Pfeffer M, Raij L, Spinosa DJ, Wilson PW; American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Kidney disease as a risk factor for development of cardiovascular disease: a statement from the American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Hypertension. 2003 Nov;42(5):1050-65. doi: 10.1161/01.HYP.0000102971.85504.7c. No abstract available. PMID 14604997
- [Background] Foley RN, Parfrey PS, Sarnak MJ. Epidemiology of cardiovascular disease in chronic renal disease. J Am Soc Nephrol. 1998 Dec;9(12 Suppl):S16-23. PMID 11443763
- [Background] Locatelli F, Marcelli D, Conte F, D'Amico M, Vecchio LD, Limido A, Malberti F, Spotti D. Survival and development of cardiovascular disease by modality of treatment in patients with end-stage renal disease. J Am Soc Nephrol. 2001 Nov;12(11):2411-2417. doi: 10.1681/ASN.V12112411. PMID 11675417
- [Background] Ok E, Asci G, Chazot C, Ozkahya M, Mees EJ. Controversies and problems of volume control and hypertension in haemodialysis. Lancet. 2016 Jul 16;388(10041):285-93. doi: 10.1016/S0140-6736(16)30389-0. Epub 2016 May 22. PMID 27226131
- [Background] Kalantar-Zadeh K, Block G, Humphreys MH, Kopple JD. Reverse epidemiology of cardiovascular risk factors in maintenance dialysis patients. Kidney Int. 2003 Mar;63(3):793-808. doi: 10.1046/j.1523-1755.2003.00803.x. PMID 12631061
- [Background] Duranti E, Imperiali P, Sasdelli M. Is hypertension a mortality risk factor in dialysis? Kidney Int Suppl. 1996 Jun;55:S173-4. PMID 8743547
- [Background] Zager PG, Nikolic J, Brown RH, Campbell MA, Hunt WC, Peterson D, Van Stone J, Levey A, Meyer KB, Klag MJ, Johnson HK, Clark E, Sadler JH, Teredesai P. "U" curve association of blood pressure and mortality in hemodialysis patients. Medical Directors of Dialysis Clinic, Inc. Kidney Int. 1998 Aug;54(2):561-9. doi: 10.1046/j.1523-1755.1998.00005.x. PMID 9690224
- [Background] Cheung AK, Sarnak MJ, Yan G, Dwyer JT, Heyka RJ, Rocco MV, Teehan BP, Levey AS. Atherosclerotic cardiovascular disease risks in chronic hemodialysis patients. Kidney Int. 2000 Jul;58(1):353-62. doi: 10.1046/j.1523-1755.2000.00173.x. PMID 10886582
- [Background] Agarwal R. Blood pressure and mortality among hemodialysis patients. Hypertension. 2010 Mar;55(3):762-8. doi: 10.1161/HYPERTENSIONAHA.109.144899. Epub 2010 Jan 18. PMID 20083728
- [Background] Kovesdy CP, Bleyer AJ, Molnar MZ, Ma JZ, Sim JJ, Cushman WC, Quarles LD, Kalantar-Zadeh K. Blood pressure and mortality in U.S. veterans with chronic kidney disease: a cohort study. Ann Intern Med. 2013 Aug 20;159(4):233-42. doi: 10.7326/0003-4819-159-4-201308200-00004. PMID 24026256
- [Background] Robinson BM, Tong L, Zhang J, Wolfe RA, Goodkin DA, Greenwood RN, Kerr PG, Morgenstern H, Li Y, Pisoni RL, Saran R, Tentori F, Akizawa T, Fukuhara S, Port FK. Blood pressure levels and mortality risk among hemodialysis patients in the Dialysis Outcomes and Practice Patterns Study. Kidney Int. 2012 Sep;82(5):570-80. doi: 10.1038/ki.2012.136. Epub 2012 Jun 20. PMID 22718187
- [Background] Port FK, Hulbert-Shearon TE, Wolfe RA, Bloembergen WE, Golper TA, Agodoa LY, Young EW. Predialysis blood pressure and mortality risk in a national sample of maintenance hemodialysis patients. Am J Kidney Dis. 1999 Mar;33(3):507-17. doi: 10.1016/s0272-6386(99)70188-5. PMID 10070915
- [Result] Bansal N, Glidden DV, Mehrotra R, Townsend RR, Cohen J, Linke L, Palad F, Larson H, Hsu CY. Treating Home Versus Predialysis Blood Pressure Among In-Center Hemodialysis Patients: A Pilot Randomized Trial. Am J Kidney Dis. 2021 Jan;77(1):12-22. doi: 10.1053/j.ajkd.2020.06.014. Epub 2020 Aug 13. PMID 32800842

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Systolic Blood Pressure (SBP) <140 mmHg: Participants will be asked to take morning and evening blood pressures every two weeks on a non-dialysis day.
  Participants will be asked to transmit these measures to the study team at minimum every 2 weeks either via Bluetooth technology, a manual log, telephone call, text message, e-mail, or verbal communication.
  Assigned intervention will be dry weight adjustment and/or adjustment of standard anti-hypertensive medications.
  Anti-Hypertensive medications: Use of standard Anti-Hypertensive medications
  Dry Weight Adjustment: The participant's target post-dialysis dry weight is adjusted
- Pre-dialysis SBP <140 mmHg: Blood pressures taken in the clinical setting at prior to start of dialysis treatment will be recorded.
  Assigned intervention will be dry weight adjustment and/or adjustment of standard anti-hypertensive medications.
  Anti-Hypertensive medications: Use of standard Anti-Hypertensive medications
  Dry Weight Adjustment: The participant's target post-dialysis dry weight is adjusted
Period: Overall Study
Arm/Group | Home Systolic Blood Pressure (SBP) <140 mmHg | Pre-dialysis SBP <140 mmHg
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — Withdrawal due to transplant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Systolic Blood Pressure (SBP) <140 mmHg | Pre-dialysis SBP <140 mmHg | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (13.1) | 56.9 (14.4) | 56.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 13 | 17 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 11 | 9 | 20
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Screen:Enrollment Ratio
Description: Percentage of eligible participants screened and eventually enrolled in the study
Time Frame: Screening
Measure: Count of Participants; unit: Participants
Groups:
- Participants Screened: Prescreened (through EMR and/or contact with nephrologists) and approached for participation in the study.
Arm/Group | Participants Screened
Number analyzed (Participants) | 70
Participants | 50

2. Primary Outcome: Adherence to Assigned Treatment Arm
Description: Percentage of participants in the home blood pressure (BP) arm who are able to measure home BP and transmit readings to the research team. Overall, across 16 wks.
Time Frame: 4 months
Population: Only the home systolic blood pressure group tested blood pressure at home
Measure: Number; unit: percentage of participants
Arm/Group | Home Systolic Blood Pressure (SBP) <140 mmHg
Number analyzed (Participants) | 25
percentage of participants
  0 BP Readings | 3
  1 BP Reading | 4
  2 BP Readings | 93

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: 1. Postdialysis unit systolic BP <90 mmHg
  2. Postdialysis unit systolic BP >200 mmHg
  3. Cramping during dialysis
  4. Syncope episodes
  5. Episodes of fall
  6. Episodes of flash pulmonary edema
  7. Symptoms of dizziness
Time Frame: Assessed every 2 weeks over 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Home Systolic Blood Pressure (SBP) <140 mmHg | Pre-dialysis SBP <140 mmHg
Number analyzed (Participants) | 25 | 25
Participants
  Postdialysis unit systolic BP <90 mmHg | 2 | 0
  Postdialysis unit systolic BP >200 mmHg | 3 | 2
  Cramping during dialysis | 13 | 18
  Syncope episodes | 1 | 1
  Episodes of fall | 3 | 6
  Episodes of flash pulmonary edema | 0 | 0
  Symptoms of dizziness | 10 | 14

4. Primary Outcome: Mean Duration (in Minutes) of Recovery From Dialysis Treatments
Description: Data were reported at study visits every 2 wks, the mean was calculated from the first to the last follow-up visit. The mean was calculated for each participant, then the overall mean was calculated for each arm.
Time Frame: Assessed every 2 weeks; Data averaged over 16 weeks
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Home Systolic Blood Pressure (SBP) <140 mmHg | Pre-dialysis SBP <140 mmHg
Number analyzed (Participants) | 25 | 25
Minutes | 327 (42) | 268 (37)

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Dialysis SBP <140 mmHg: Blood pressures taken in the clinical setting at prior to start of dialysis treatment will be recorded.
  Assigned intervention will be dry weight adjustment and/or adjustment of standard anti-hypertensive medications.
  Anti-Hypertensive medications: Use of standard Anti-Hypertensive medications
  Dry Weight Adjustment: The participant's target post-dialysis dry weight is adjusted
Arm/Group | Home Systolic Blood Pressure (SBP) <140 mmHg | Dialysis SBP <140 mmHg
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/25
Other Adverse Events (participants affected / at risk) | 25/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Home Systolic Blood Pressure (SBP) <140 mmHg (N=25) | Dialysis SBP <140 mmHg (N=25)
Syncope (Cardiac disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Home Systolic Blood Pressure (SBP) <140 mmHg (N=25) | Dialysis SBP <140 mmHg (N=25)
Fall (General disorders) | 3 | 6
Cramping (Musculoskeletal and connective tissue disorders) | 13 | 18
Symptoms of dizziness (General disorders) | 10 | 14
Symptoms of lightheadedness (General disorders) | 14 | 12
Predialysis SBP < 90 mm Hg (Cardiac disorders) | 1 | 2
Postdialysis SBP < 90 mm Hg (Cardiac disorders) | 2 | 0
Predialysis SBP > 200 mm Hg (Cardiac disorders) | 4 | 4
Postdialysis SBP > 200 mm Hg (Cardiac disorders) | 3 | 2
Symptoms of fatigue (General disorders) | 15 | 16
Intradialytic hypotension (Cardiac disorders) | 21 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03459807/Prot_SAP_001.pdf
  • Informed Consent Form (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03459807/ICF_002.pdf